CLINICAL TRIAL: NCT04662307
Title: An Intelligent Cardiopulmonary Rehabilitative System on Cardiopulmonary Fitness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Director of Physical Medicine and Rehabilitation, Taipei Medical University WanFang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N202005081
Record Dates: First submitted 2020-11-25; First posted 2020-12-10 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Lifestyle, Sedentary
Keywords: cardiac rehabilitation; cardiorespiratory fitness; aerobic exercise; endurance training
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A small group of healthy subjects with sedentary lifestyle is recruited to validate the ICRS. They receive training with ICRS three sessions a week, for a total of 12 sessions. The outcome assessments are performed before and after the training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intelligent cardiopulmonary rehabilitation system (ICRS) (Experimental): The intelligent cardiopulmonary rehabilitation system is designed to improve the user's adherence to pre-determined training intensity. The training intensity is pre-determined using the 60%-80% heart rate reserve which is obtained from the cardiopulmonary exercise test at prestest. The system allows dynamically auto-adjust the paddling resistance in accordance to the patient's current hear rate and paddling rate, with the goal to maintain the patient's heart rate at the pre-determined heart rate zone through the training period.
  Interventions: Device: Intelligent cardiopulmonary rehabilitation system (ICRS)

INTERVENTIONS:
Device: Intelligent cardiopulmonary rehabilitation system (ICRS) — Participants are required to wear a wristband heart rate monitor and exercise on a cycling ergometer-based ICRS for 30 minutes (5 minute of warm-up, 20 minutes of training followed by 5 minutes of cooldown). The target intensity for the 20-min training period is set at 60%~80% HRR determined in the pretest of cardiopulmonary exercise test.

SUMMARY:
Contemporary cardiopulmonary rehabilitation programs often utilize cycling ergometer, involving one-on-one heart rate monitoring by physiotherapists to ensure that patients reach the target training intensity during training sessions. However, the process is frequently described as monotonous and boring, resulting in early fatigue of therapists and patients as well as poor compliance, leading to undertraining and suboptimal outcomes.

This study aims to test the feasibility of the "Intelligent Cardiopulmonary Training System (ICRS)" and a novel indicator of measuring the adherence to training intensity. The ICRS was developed with the idea to provide machine-based supervision on the user's heart rate during training. It provides moderate-intensity continuous training with a cycling ergometer. This system automatically adjusts the paddling resistance according to the user's real-time heart rate, and helps to improve the user's adherence to pre-determined training intensity without trainer's watch. The automation of intensity adjustment has its potential for conditions in which supervision is not feasible.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary healthy people

Exclusion Criteria:

* Patients whose heart rate can not be used as the indicator of training intensity (eg, ar-rhythmia, atrial fibrillation, beta-blockers users)
* With any reason that the patient is not suitable to undergo
* Patients who are unable to do cycling due to musculoskeletal problems
* Patients who can not follow the instruction of trainers due to cognitive or emotional-problems.
* Patients whose medical condition is not unstable.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2-peak) | 4 weeks
  Peak oxygen consumption is measured by cardiopulmonary test.

SECONDARY OUTCOMES:
Peak workload | 4 weeks
  Peak workload is measured by cardiopulmonary exercise test
percentage of time (%time) within the pre-determined target heart rate | 4 weeks
  The ICRS outputs the heart rate-time plots and calculated the %time for each session

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Nung Lin, MD, Principal Investigator — Wan-Fang Hospital, Taipei Medical University
Locations (1):
- Department of rehabilitation, WanFang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No